CLINICAL TRIAL: NCT04668092
Title: Immediate Effects of Functional Dry Needling on the Length of Shortened Hamstring Muscle
Brief Title: Functional DN for Shortened HS Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/00767 Qaisar Ali Khan
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Hamstring Contractures
Keywords: Dry needling; LEFS; 90-90 SLR

STUDY DESIGN:
Masking Description: assessor who helped to record the measurement was blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional dry needling (Experimental): Functional dry needling for shortened hamstring muscle
  Interventions: Other: Functional dry needling

INTERVENTIONS:
Other: Functional dry needling — functional dry needling applied to hamstring for 1 minute and post interventional data collected

SUMMARY:
The aim of this study is to find whether functional dry needle is helpful to increase the length of shortened hamstring muscle or not

DETAILED DESCRIPTION:
Single pretest-post clinical trial to find immediate effects of functional dry needling to increase the length of the shortened hamstring. This study will be carried on single group which will include male subjects only. The data will be recorded before and immediately after the treatment. A monofilament stainless steel needle will be inserted on three points on hamstring muscle which will include semitendinosus, semimembranosus and bicep femoris. Treatment session will consist of 1 minute 20 seconds for each point on the hamstring and the manipulation will be performed by "Pistoning technique" in which the needle will be drawn out (not fully out of skin) after inserted and then again pushed in and data will be recorded after the treatment session on the basis of increase in length of hamstring which will be measure through 90-90 SLR (AKE) and on the lower extremity functional scale (LEFS)

ELIGIBILITY:
Inclusion Criteria:

* Having hamstring length less than 80 degree during 90-90 SLR on goniometer,
* also the subject that suffers from knee Osteoarthritis,
* Spondylosis,
* LBP,
* Lumber radiculopathy,
* Subjects with MTrPs and those with hyper lordosis were recruited in the study

Exclusion Criteria:

* subjects suffering from blood clotting disorders such as hemophilia,
* those with deformities such as leg length discrepancy,
* compromised immune system,
* vascular diseases,
* Diabetes,
* People with congenital or metabolic bone disease such as Spondyloepiphyseal Dysplasia and Pregnancy were excluded from the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
90-90 Straight Leg Raise (SLR) | 1 day
  90-90 Straight Leg Raise (SLR) test is used to measure hamstring length through goniometer. The patient lie supine and flex the hip and extend the knee. The test is positive if the patient cannot go withing last 20 degrees of knee extension.

SECONDARY OUTCOMES:
Lower extremity Functional scale (LEFS) | 1 day
  Lower extremity Functional Scale is a 20 content scale design to measure the disability level of the patient on the basis of function of the lower extremity. Score ranges from "0" to "80". The lower the score the greater is the disability.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Saidu group of teaching hospital said sharif swat, Swat, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Adkitte R, Rane SG, Yeole U, Nandi B, Gawali P. Effect of muscle energy technique on flexibility of hamstring muscle in Indian national football players. Saudi Journal of Sports Medicine. 2016;16(1):28. — https://scholar.google.com/
- See also: Odunaiya N, Hamzat T, Ajayi O. The effects of static stretch duration on the flexibility of hamstring muscles. African journal of biomedical research. 2005;8(2):79-82. — https://scholar.google.com/
- See also: Phrompaet S, Paungmali A, Pirunsan U, Sitilertpisan P. Effects of pilates training on lumbo-pelvic stability and flexibility. Asian Journal of sports medicine. 2011;2(1):16. — https://scholar.google.com/
- See also: Wang SS, Whitney SL, Burdett RG, Janosky JE. Lower extremity muscular flexibility in long distance runners. Journal of Orthopaedic & Sports Physical Therapy. 1993;17(2):102-7. — https://scholar.google.com/
- See also: Akinpelu AO, Bakare U, Adegoke BA. Influence of age on hamstring tightness in apparently healthy Nigerians. Journal of Nigeria Society of Physiotherapy. 2009;15(2):35-41. — https://scholar.google.com/
- See also: Cagnie B, Elliott J, O'Leary S, D'hooge R, Dickx N, Danneels L. Muscle functional MRI as an imaging tool to evaluate muscle activity. journal of orthopaedic & sports physical therapy. 2011;41(11):896-903 — https://scholar.google.com/
- See also: Hidler JM, Rymer WZ. A simulation study of reflex instability in spasticity: origins of clonus. IEEE Transactions on Rehabilitation Engineering. 1999;7(3):327-40 — https://scholar.google.com/
- See also: Lance JW. Pathophysiology of spasticity and clinical experience with baclofen. Spasticity: disordered motor control. 1980:185-204. — https://scholar.google.com/
- See also: Waseem M, Nuhmani S, Ram C. Efficacy of Muscle Energy Technique on hamstring muscles flexibility in normal Indian collegiate males. Calicut medical journal. 2009;7(2):e4. — https://scholar.google.com/
- See also: Smith LR, Chambers HG, Subramaniam S, Lieber RL. Transcriptional abnormalities of hamstring muscle contractures in children with cerebral palsy. PloS one. 2012;7(8):e40686. — https://scholar.google.com/
- See also: Smith LR. Skeletal muscle adaptations in hamstring contractures of children with cerebral palsy: UC San Diego; 2011. — https://scholar.google.com/
- See also: Jóźwiak M, Pietrzak S, Tobjasz F. The epidemiology and clinical manifestations of hamstring muscle and plantar foot flexor shortening. Developmental Medicine & Child Neurology. 1997;39(7):481-3. — https://scholar.google.com/
- See also: Erkula G, Demirkan F, Kılıç BA, Kıter E. Hamstring shortening in healthy adults. Journal of Back and Musculoskeletal Rehabilitation. 2002;16:77-81. — https://scholar.google.com/
- See also: Klotz MC, Hirsch K, Heitzmann D, Maier MW, Hagmann S, Dreher T. Distal femoral extension and shortening osteotomy as a part of multilevel surgery in children with cerebral palsy. World Journal of Pediatrics. 2017;13(4):353-9. — https://scholar.google.com/
- See also: H, Garrett WE, Moorman CT, Yu B. Injury rate, mechanism, and risk factors of hamstring strain injuries in sports: a review of the literature. Journal of sport and health science. 2012;1(2):92-101. — https://scholar.google.com/
- See also: Askling C, Lund H, Saartok T, Thorstensson A. Self-reported hamstring injuries in student-dancers. Scandinavian journal of medicine & science in sports. 2002;12(4):230-5 — https://scholar.google.com/
- See also: Bron C, Dommerholt JD. Etiology of myofascial trigger points. Current pain and headache reports. 2012;16(5):439-44. — https://scholar.google.com/
- See also: rophy RH, Chehab EL, Barnes RP, Lyman S, Rodeo SA, Warren RF. Predictive value of orthopedic evaluation and injury history at the NFL combine. Medicine and science in sports and exercise. 2008;40(8):1368-72. — https://scholar.google.com/
- See also: Woods C, Hawkins R, Hulse M, Hodson A. The Football Association Medical Research Programme: an audit of injuries in professional football-analysis of preseason injuries. British journal of sports medicine. 2002;36(6):436-41. — https://scholar.google.com/
- See also: lmer EB, Wenger DR, Mubarak SJ, Sutherland DH. Proximal hamstring lengthening in the sitting cerebral palsy patient. Journal of pediatric orthopedics. 1992;12(3):329-36. — https://scholar.google.com/
- See also: Hess T, Gleitz M, Egert S, Hopf T. Chondropathia patellae and knee muscle control. Archives of orthopaedic and trauma surgery. 1996;115(2):85-9. — https://scholar.google.com/
- See also: Hoffinger SA, Rab GT, Abou-Ghaida H. Hamstrings in cerebral palsy crouch gait. Journal of pediatric orthopedics. 1993;13(6):722-6. — https://scholar.google.com/
- See also: Papagelopoulos PJ, Sim FH. Patellofemoral pain syndrome: diagnosis and management. Orthopedics. 1997;20(2):148-57. — https://scholar.google.com/
- See also: Lin JP, Brown JK, Brotherstone R. Assessment of spasticity in hemiplegic cerebral palsy. II: Distal lower-limb reflex excitability and function. Developmental Medicine & Child Neurology. 1994;36(4):290-303. — https://scholar.google.com/
- See also: Baker RT, Hansberger BL, Warren L, Nasypany A. A novel approach for the reversal of chronic apparent hamstring tightness: a case report. International journal of sports physical therapy. 2015;10(5):723. — https://scholar.google.com/
- See also: Hosman AJ, de Kleuver M, Anderson PG, van Limbeek J, Langeloo DD, Veth RP, et al. Scheuermann kyphosis: the importance of tight hamstrings in the surgical correction. Spine. 2003;28(19):2252-9. — https://scholar.google.com/
- See also: Smith JA, Hu SS. Management of spondylolysis and spondylolisthesis in the pediatric and adolescent population. Orthopedic Clinics of North America. 1999;30(3):487-99. — https://scholar.google.com/
- See also: Sheptak PE, Susen AF. Diastematomyelia. American Journal of Diseases of Children. 1967;113(2):210-3. — https://scholar.google.com/
- See also: Zurakowski D, Kriemler S, Micheli LJ. Spondylolysis: returning the athlete to sports participation with brace treatment. Orthopedics. 2002;25(6):653-7. — https://scholar.google.com/